CLINICAL TRIAL: NCT01167621
Title: Assessment of Extravascular Lung Water and Hemodynamics Changes in Patients Treated by High Frequency Oscillation-ventilation for Refractory ARDS
Brief Title: Changes in Refractory Acute Respiratory Distress Syndrome (ARDS) Patients Under High Frequency Oscillation-ventilation
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/CHR/01
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Refractory Acute Respiratory Distress Syndrome; Indexed Extra-vascular Lung Water; HFO-ventilation
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study is intended to evaluate the hemodynamic and the indexed extrapulmonary lung water (ELWI) changes in patients treated by high frequency oscillation-ventilation (HFO-V) for refractory acute respiratory distress syndrome (ARDS). HFO-V may be used as rescue treatment in refractory ARDS but its hemodynamic impact is discussed. Moreover, as Extra Vascular Lung Water (a transpulmonary thermodilution parameter) was proven to be an independent mortality factor in ICU-patients, the investigators decided to monitor it in all ARDS patients who ended up needing HFO-V, from HFO-V plugging under 72 hours of this type of ventilation. All ARDS patients underwent high Positive End Expiratory Pressure (PEEP) with "protective ventilation" and those who remained below a PaO2/FiO2 ratio of 120 after 24h will be considered as "refractory ARDS patients" and, therefore eligible. They will be monitored by the transpulmonary thermodilution PiCCO technique (Pulsion Medical System. Munich, Germany) and placed under HFO-V. Both transpulmonary thermodilution measurements (ELWI , Cardiac Output, Global End-diastolic Volume) and standard transthoracic echocardiographic measurements (Ejection Fraction, End-diastolic Right and Left Ventricular Area, preload indexes) were be performed from HFO-V plugging to Day 3. The investigators suggest that ELWI will be correlated to HFO-V responsiveness and that cardiac output will not change at the HFO-V plugging, regardless of preload indexes variation. Inclusion will be proceeded over a 2 year period and, according to the population, the investigators expect about 50 eligible patients.

DETAILED DESCRIPTION:
All ARDS patients will be treated according to a strictly defined protocol. Each patient will receive a standardised sedation with sufentanil, midazolam and atracurium. Tidal volume was adjusted on 6ml/kg of ideal body weight based on the height of each patient. Positive End Expiratory Pressure (PEEP) will be settled at the highest possible level (from 5 to 18cmH2O) without exceeding a plateau pressure below 30cmH2O. The oxygenation goal will a pulse oximeter saturation above 88%. Ventilation parameters will be adapted to the results of arterial blood gas samples realised 3 times a day.

Refractory patients will be defined by a PaO2/FiO2 ratio below 120 and will be eligible for "rescue techniques" like HFOV, prone position, nitrous oxide, Extra Corporeal Membrane Oxygenation (ECMO). Clinician choice for each technique will be unguided but if any rescue technique will be used prior to HFOV, patient will be not eligible for the study. All the patients will be monitored by a transpulmonary PiCCO technique. In every case, a femoral artery catheter (20cm, 5 French Pulsiocath, Pulsion Medical System) will be used for recording pressure and thermodilution signals via the PiCCOplus device V6.0 (Pulsion Medical System, Munich, Germany) using a venous central catheter.

Patients meeting the inclusion criteria after 12h of standardised ventilation will be placed under HFO-V and closely monitored by arterial blood gas sample, PiCCO-derived measurements and transthoracic echocardiography (primary and secondary outcome measures detailed later on).

HFOV failure will be defined by PaO2/FiO2<70 or hypercapnia > 55mmHg after optimisation of the HFO-V settings. In case of HFO-V failure, nitrous oxide will be used in first place as a complementary technique. In case of inefficacy, the investigators would switch to any other technique, causing the exclusion of the protocol.

HFOV weaning technique is also standardised : FiO2 will be lowered gradually 10 percents by 10 percents until 40% is reached. Then, the mean pressure will follow the same gradual lowering (2cmH2O by 2cmH2O until 24cmH2O). Once these two thresholds are reached, a HFOV weaning attempt will be realised with standard ventilation.

The investigators will also report any therapeutics that may influence hemodynamic measurements such as fluid challenge, diuretics, norepinephrine and sedation.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Admission in ICU
* Transpulmonary PiCCO-technique monitoring
* Refractory ARDS (ratio PaO2/FiO2 < 120) after 12 hours of protective mechanical ventilation with maximal PEEP recruitment (inclusion is possible before this 12hours delay if the patient's status is worsening under optimised ventilation parameters AND plateau pressure above 30cm H2O OR saturation <88%)
* Choice of HFO-V as ventilation rescue technique
* Hemodynamic stability at plugging (after fluid challenge or norepinephrine if necessary)

Exclusion Criteria:

* Arteritis, hemostasis disorder
* Pneumothorax,
* Acute cardiac failure indicating a ECLS
* Previous use of other rescue techniques (Nitrous oxide, prone ventilation, ECMO)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Refractory Acute Respiratory Distress Syndrome (ARDS) patients admitted to the Intensive Care Unit of Saint-Denis hospital (REUNION ISLAND)
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Indexed Extra Vascular Lung Water (EVLWI) changes under HFO ventilation | 3-day period after HFO-V

SECONDARY OUTCOMES:
Hemodynamics changes under HFO ventilation | 3-day period after HFO-V

CONTACTS AND LOCATIONS:
Overall Officials: Julien Jabot, MD, Principal Investigator — University Hospital Reunion Island - Felix Guyon Site
Locations (1):
- Réanimation polyvalente, University Hospital Reunion Island - Felix Guyon Site, Saint Denis de La Réunion, France

REFERENCES:
- [Background] Simma B, Fritz M, Fink C, Hammerer I. Conventional ventilation versus high-frequency oscillation: hemodynamic effects in newborn babies. Crit Care Med. 2000 Jan;28(1):227-31. doi: 10.1097/00003246-200001000-00038. PMID 10667528
- [Background] Traverse JH, Korvenranta H, Adams EM, Goldthwait DA, Carlo WA. Cardiovascular effects of high-frequency oscillatory and jet ventilation. Chest. 1989 Dec;96(6):1400-4. doi: 10.1378/chest.96.6.1400. PMID 2684557
- [Background] Arnold JH, Truog RD, Thompson JE, Fackler JC. High-frequency oscillatory ventilation in pediatric respiratory failure. Crit Care Med. 1993 Feb;21(2):272-8. doi: 10.1097/00003246-199302000-00021. PMID 8428481
- [Background] Zobel G, Dacar D, Rodl S. Hemodynamic effects of different modes of mechanical ventilation in acute cardiac and pulmonary failure: an experimental study. Crit Care Med. 1994 Oct;22(10):1624-30. PMID 7924375
- [Background] Jabot J, Teboul JL, Richard C, Monnet X. Passive leg raising for predicting fluid responsiveness: importance of the postural change. Intensive Care Med. 2009 Jan;35(1):85-90. doi: 10.1007/s00134-008-1293-3. Epub 2008 Sep 16. PMID 18795254
- [Background] Monnet X, Osman D, Ridel C, Lamia B, Richard C, Teboul JL. Predicting volume responsiveness by using the end-expiratory occlusion in mechanically ventilated intensive care unit patients. Crit Care Med. 2009 Mar;37(3):951-6. doi: 10.1097/CCM.0b013e3181968fe1. PMID 19237902
- [Background] Sakka SG, Klein M, Reinhart K, Meier-Hellmann A. Prognostic value of extravascular lung water in critically ill patients. Chest. 2002 Dec;122(6):2080-6. doi: 10.1378/chest.122.6.2080. PMID 12475851
- [Background] Craig TR, Duffy MJ, Shyamsundar M, McDowell C, McLaughlin B, Elborn JS, McAuley DF. Extravascular lung water indexed to predicted body weight is a novel predictor of intensive care unit mortality in patients with acute lung injury. Crit Care Med. 2010 Jan;38(1):114-20. doi: 10.1097/CCM.0b013e3181b43050. PMID 19789451
- [Background] Mercat A, Richard JC, Vielle B, Jaber S, Osman D, Diehl JL, Lefrant JY, Prat G, Richecoeur J, Nieszkowska A, Gervais C, Baudot J, Bouadma L, Brochard L; Expiratory Pressure (Express) Study Group. Positive end-expiratory pressure setting in adults with acute lung injury and acute respiratory distress syndrome: a randomized controlled trial. JAMA. 2008 Feb 13;299(6):646-55. doi: 10.1001/jama.299.6.646. PMID 18270353
- [Derived] Ursulet L, Roussiaux A, Belcour D, Ferdynus C, Gauzere BA, Vandroux D, Jabot J. Right over left ventricular end-diastolic area relevance to predict hemodynamic intolerance of high-frequency oscillatory ventilation in patients with severe ARDS. Ann Intensive Care. 2015 Dec;5(1):25. doi: 10.1186/s13613-015-0068-6. Epub 2015 Sep 17. PMID 26380993